CLINICAL TRIAL: NCT05767554
Title: Depression, Experiential Diversity, and Behavioral Novelty: A Mobile Sensing Experimental Paradigm
Brief Title: Depression, Experiential Diversity, and Behavioral Novelty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Christopher G. Beevers, Professor of Psychology, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003773
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Depression
Keywords: Behavioral activation; Mobile sensing
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief modified behavioral activation (Experimental): Participants randomized to the behavioral activation condition will meet with a graduate level clinician for one hour.
  Interventions: Behavioral: Brief modified behavioral activation
- Measurement-only control (No Intervention): Participants who are not randomized to the active condition will take part in a measurement-only control condition. They will participate in all portions of the study except for the in-person behavioral activation session. They will complete a baseline and fill out daily surveys.

INTERVENTIONS:
Behavioral: Brief modified behavioral activation — The clinician will deliver psychoeducation about the nature of depression and the rationale behind the behavioral activation model (i.e. increasing level of activation can begin a positive feedback cycle of reward and improvements in mood state). Participants will be encouraged to add new, enjoyable activities to their daily schedules. Clinicians will emphasize the importance of novelty and increased engagement with the surrounding environment in the psychoeducational portion and in activity scheduling.
  Arms: Brief modified behavioral activation

SUMMARY:
The purpose of the study is to test whether changes in behavioral patterns are related to changes in depression. Depression is a psychological condition that involves persistent sad mood and/or an inability to enjoy pleasurable activities. Very stable behavioral patterns may be related to symptoms of depression. The aim of this study is to learn more about the relationship between symptoms of depression and behavioral patterns that are collected via global positioning system location data from a smart phone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Possession and daily use of a smart phone
* Able to speak and read English
* Patient Health Questionnaire -8 (PHQ-8) > 10
* Behavioral Activation for Depression (BADS) Activation Subscale < 16
* Ability to complete all study procedures

Exclusion Criteria:

* Self-reported lifetime diagnosis of agoraphobia or bipolar disorder
* Severe neurodevelopmental disorder
* Major travel plans within study period

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-8 Total Score over 5 Weeks | Baseline and 5 weeks
  Level of depression symptoms assessed weekly by the Patient Health Questionnaire - 8 via smart phone survey. The PHQ-8 ranges from 0-24 with higher scores indicating more severe symptoms of depression.

SECONDARY OUTCOMES:
Change in Behavioral Activation for Depression Scale over 5 Weeks | Baseline and 5 weeks
  Level of behavioral activation as measured by the Behavioral Activation for Depression Scale (BADS). The BADS ranges from 0-150 with higher scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Beevers, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin Institute of Mental Health Research, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No